CLINICAL TRIAL: NCT03495791
Title: Web (YouTube) Based Educational Intervention to Improve Patient-Physician Awareness of Cardiovascular Risk in Rheumatoid Arthritis.
Brief Title: Educational Intervention to Improve Patient-Physician Awareness of Cardiovascular Risk in Rheumatoid Arthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14090405
Record Dates: First submitted 2018-03-14; First posted 2018-04-12 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Arthritis, Rheumatoid
Keywords: RA; Rheumatoid Arthritis; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EI development phase. (Experimental)
  Interventions: Other: YouTube Video
- Pilot-testing phase. (No Intervention)

INTERVENTIONS:
Other: YouTube Video — Educational Video
  Arms: EI development phase.

SUMMARY:
This study will provide an educational intervention through means of a video to educate subjects on the risk of cardiovascular health on Rheumatoid arthritis.

DETAILED DESCRIPTION:
Subjects will be randomized into an interventional group and non-interventional group. Both groups will perform several surveys before an educational intervention may be given. Both Groups will come back 3 months post visit to complete additional surveys.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnoses of Rheumatoid Arthritis of at least 3 months by a Rheumatologist

Exclusion Criteria:

* Inability to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Heart Disease Knowledge Questionnaire | 3 Months
  30 items survey completed at baseline (pre-intervention, post intervention), and 3 month follow-up. Change in cardiovascular knowledge at 3 months and baseline (post-intervention) will be measured against baseline pre-intervention values.
Heart Disease Fact Questionnaire | 3 Months
  13 items survey completed at baseline (pre-intervention, post intervention), and 3 month follow-up. Change in cardiovascular awareness at 3 months and baseline (post-intervention) will be measured against baseline pre-intervention values.

SECONDARY OUTCOMES:
Statues of Hyperlipidemia treatment | 1 Year
  Change in hyperlipidemia treatment from Screening to 1 year.
Cholesterol | 1 year
  Change in Cholesterol from Screening to 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

DOCUMENTS (1):
  • Study Protocol (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03495791/Prot_000.pdf